CLINICAL TRIAL: NCT00486902
Title: Does a Single Intravenous Dose of Ketamine Reduce the Need for Supplemental Opioids in Post-Cesarean Section Patients?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0524-030
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Ketamine Adverse Reaction; Effects of; Anesthesia, Spinal and Epidural, in Pregnancy; Complication of Labor and/or Delivery
Keywords: Ketamine; Spinal Anesthesia; C-section
MeSH Terms: interventions — Ketamine; N-Methylaspartate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Subjects receive IV ketamine 10 mg 5 minutes after infant delivery.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Subjects receive IV Saline 20 mL 5 minutes after infant delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Ketamine 10 mg diluted to 20 mL delivered over 10 minutes via an infusion pump set at 2ml/minute
  Other Names: N-methyl-D-aspartate (NMDA)
  Arms: Ketamine
Drug: Placebo — Saline 20 mL IV infusion delivered over 10 minutes via an infusion pump set at 2ml/minute
  Other Names: 0.9% Saline
  Arms: Placebo

SUMMARY:
Pain control after cesarean delivery is associated with improved breastfeeding and infant rooming-in times. In addition, inadequate analgesia leads to elevated plasma catecholamine concentrations, which negatively affect every organ system. There is growing evidence that ketamine, N-methyl-D-aspartate receptor antagonist, is efficacious when used as an adjuvant in postoperative pain control. A 2006 Cochrane Collaboration systemic review and meta-analysis concluded, "Ketamine in subanesthetic doses….is effective in reducing morphine requirements in the first 24 hours after surgery."

Ketamine's prolonged analgesic effect, despite its short half-life and its use in low doses, is theorized to be due to blockade of spinal cord central sensitization. Central sensitization is a phenomenon whereby repeated painful stimulus leads to more severe pain perception over time despite no change in the intensity of the painful stimulus.Ketamine may also prevent the development of acute opioid tolerance. Ketamine's analgesic effects have also demonstrated in the obstetric population. Post-cesarean delivery morphine requirements in women who received ketamine as part of a general anesthesia technique were decreased. Similary, low-dose ketamine in conjunction with bupivacaine-only spinal anesthesia reduced postoperative analgesic requirements compared to bupivacaine-only spinal anesthesia and bupivacaine-fentanyl spinal anesthesia.

In the United States, healthy women scheduled for elective cesarean delivery commonly receive spinal anesthesia with bupivacaine-fentanyl-morphine. To our knowledge, IV ketamine has not been studied as an adjuvant to this regimen in the analgesic management in post-cesarean delivery patients. Multimodal therapy for postoperative pain control is widely practiced due to the advantage it provides in blocking multiple pain pathways while minimizing side effects of each individual pain medication. We hypothesize that low dose intravenous ketamine will improve multi-modal post-cesarean analgesia compared to placebo. The purpose of this study is to evaluate this hypothesis and study the possible side effects of this regimen in combination with bupivacaine-fentanyl-morphine spinal anesthesia.

DETAILED DESCRIPTION:
Eligible women for elective cesarean section admitted to the Labor and Delivery Unit of Prentice Women's Hospital will be approached for study participation immediately after the routine preanesthetic evaluation. This occurs shortly after admission to the Labor and Delivery Unit. Women who agree to participate will give written, informed consent at this time.

Subjects will be prepared preoperatively in the usual fashion with intravenous (IV) access, aspiration prophylaxis and intraoperative monitoring. Preincision antibiotics will be given and uterotonic medications will be used as per usual practice after delivery.

The anesthesiologist will perform a spinal anesthetic per routine with the subject in the sitting position using sterile technique at the L3-4 interspace (± one vertebral interspace). The spinal anesthetic will consist of 12 mg of hyperbaric bupivacaine + 15 μg fentanyl + 150 μg of morphine. The subject will be placed supine with left lateral tilt to alleviate aortocaval compression. Cesarean section will commence after adequate anesthesia is assured to a T4 sensory level to pinprick. Vasopressors and IV fluids will be administered at the anesthesiologist's discretion per usual practice.

At the time of delivery, subjects will be randomized to one of two groups using a computer generated random number table. Randomization will be blocked based on whether the cesarean procedure is a primary or a repeat procedure. Randomization assignments will be kept in sequentially numbered opaque envelopes. The envelope will be opened by a research nurse who will prepare a 20 mL syringe labeled "study drug". The syringe will be given to the anesthesiologist blinded to the treatment group who will subsequently administer the study drug. Subjects randomized to the treatment group will receive ketamine 10 mg (ketamine 10 mg/mL) diluted to 20 mL with 0.9% preservative free saline. Subjects randomized to the placebo group will receive 20 mL preservative free saline.

The study drug will be administered into the intravenous line via an infusion pump over 10 minutes. Five minutes after placebo or drug administration, the anesthesiologist will ask the subject if she has nausea, vomiting and pruritus. Nausea and pruritus will be graded as none, mild, moderate or severe; and vomiting as present or absent. Any spontaneous complaints of psychedelic effects will be noted at this time. Sedation will be assessed via the Richmond agitation-sedation scale (RASS [see Appendix 1]).

Upon completion of the cesarean section, the subject will be transported to the post anesthesia recovery unit. Patients will receive ketorolac 30 mg every 6 hours time 4 doses beginning shortly after admission to the PACU.

At 1 h, 4 h, 8 h, 12 h and at 24 h after administration of the study drug, the subject's pain will be assessed using the numeric rating scale for pain NRS 0-10 (see Appendix 2). Patients may request rescue analgesia if they are experiencing discomfort. The time of first rescue analgesia request will be noted, and the NRS will be determined at the time of request for rescue analgesia.

Rescue medication will consist of hydrocodone 10 mg plus acetaminophen 325 mg per os. An additional dose of hydrocodone 10 mg plus acetaminophen 325 mg will be provided after 1 hour if the pain is not relieved to the subject's satisfaction. These are routine oral analgesic medications for postoperative cesarean delivery analgesia. Standard orders will be written for monitoring sedation and respiratory rate, and treatment of side effects (nausea, vomiting, pruritus and respiratory depression). The total amount of rescue medication will be determined for each subject after 24, 48 and 72 hours.

The presence of nausea, vomiting, and pruritus will be assessed at the same time intervals as the NRS for pain: 1 h, 4 h, 8 h, 12 h and 24 h after IV infusion of ketamine or placebo. The subjective psychedelic effects of ketamine and morphine will be assessed using a set of true/false questions from the LSD and morphine short form of the Addiction Research Center Inventory, ARCI (Appendix 3). These questions will be administered verbally by the anesthesiologist or researcher blinded to the treatment group upon admission to the PACU and at 4 h.

The following data will be collected in addition to the primary and secondary outcome data: maternal age, height, weight, prepregnancy weight, gestational age and IV fluids administered during cesarean section. In addition, all intraoperative and postoperative medications will be recorded, including those administered for the treatment of side effects listed above.

Protocol specific analgesia assessment ends 24 hours after administration of the study drug. At 72 hours the subject will be asked about her satisfaction with postoperative analgesia (100 mm scale, 0 mm = not satisfied at all, 100 mm = very satisfied). One telephone follow-up evaluation 2 weeks after delivery will again, assess for satisfaction with analgesia and average pain (NRS) since the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women are at term (≥37 week gestation),
* Healthy,
* ASA class 1-2,
* Scheduled for elective cesarean section whose anesthetic plan is for spinal anesthesia with intrathecal morphine and intravenous ketorolac analgesia for post operative analgesia

Exclusion Criteria:

* Women with American Society of Anesthesiologists physical status >2,
* Body mass index ≥40 kg/m2,
* Known allergy to any of the study medications,
* Contraindication to the spinal anesthesia,
* History of substance abuse,
* History of hallucinations,
* Chronic opioid therapy,
* Chronic pain.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Yost NP, Bloom SL, Sibley MK, Lo JY, McIntire DD, Leveno KJ. A hospital-sponsored quality improvement study of pain management after cesarean delivery. Am J Obstet Gynecol. 2004 May;190(5):1341-6. doi: 10.1016/j.ajog.2003.10.707. PMID 15167840
- [Background] Subramaniam K, Subramaniam B, Steinbrook RA. Ketamine as adjuvant analgesic to opioids: a quantitative and qualitative systematic review. Anesth Analg. 2004 Aug;99(2):482-95, table of contents. doi: 10.1213/01.ANE.0000118109.12855.07. PMID 15271729
- [Background] Bell RF, Dahl JB, Moore RA, Kalso E. Perioperative ketamine for acute postoperative pain. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD004603. doi: 10.1002/14651858.CD004603.pub2. PMID 16437490
- [Background] Menigaux C, Fletcher D, Dupont X, Guignard B, Guirimand F, Chauvin M. The benefits of intraoperative small-dose ketamine on postoperative pain after anterior cruciate ligament repair. Anesth Analg. 2000 Jan;90(1):129-35. doi: 10.1097/00000539-200001000-00029. PMID 10624993
- [Background] Menigaux C, Guignard B, Fletcher D, Sessler DI, Dupont X, Chauvin M. Intraoperative small-dose ketamine enhances analgesia after outpatient knee arthroscopy. Anesth Analg. 2001 Sep;93(3):606-12. doi: 10.1097/00000539-200109000-00016. PMID 11524327
- [Background] Kwok RFK, Lim J, Chan MTV, Gin T, Chiu WKY. Preoperative ketamine improves postoperative analgesia after gynecologic laparoscopic surgery. Anesth Analg. 2004 Apr;98(4):1044-1049. doi: 10.1213/01.ANE.0000105911.66089.59. PMID 15041596
- [Background] Argiriadou H, Himmelseher S, Papagiannopoulou P, Georgiou M, Kanakoudis F, Giala M, Kochs E. Improvement of pain treatment after major abdominal surgery by intravenous S+-ketamine. Anesth Analg. 2004 May;98(5):1413-8, table of contents. doi: 10.1213/01.ane.0000111204.31815.2d. PMID 15105223
- [Background] Guillou N, Tanguy M, Seguin P, Branger B, Campion JP, Malledant Y. The effects of small-dose ketamine on morphine consumption in surgical intensive care unit patients after major abdominal surgery. Anesth Analg. 2003 Sep;97(3):843-847. doi: 10.1213/01.ANE.0000075837.67275.36. PMID 12933413
- [Background] Guignard B, Coste C, Costes H, Sessler DI, Lebrault C, Morris W, Simonnet G, Chauvin M. Supplementing desflurane-remifentanil anesthesia with small-dose ketamine reduces perioperative opioid analgesic requirements. Anesth Analg. 2002 Jul;95(1):103-8, table of contents. doi: 10.1097/00000539-200207000-00018. PMID 12088951
- [Background] Xie H, Wang X, Liu G, Wang G. Analgesic effects and pharmacokinetics of a low dose of ketamine preoperatively administered epidurally or intravenously. Clin J Pain. 2003 Sep-Oct;19(5):317-22. doi: 10.1097/00002508-200309000-00006. PMID 12966258
- [Background] Suzuki M, Tsueda K, Lansing PS, Tolan MM, Fuhrman TM, Ignacio CI, Sheppard RA. Small-dose ketamine enhances morphine-induced analgesia after outpatient surgery. Anesth Analg. 1999 Jul;89(1):98-103. doi: 10.1097/00000539-199907000-00017. PMID 10389785
- [Background] Aida S, Yamakura T, Baba H, Taga K, Fukuda S, Shimoji K. Preemptive analgesia by intravenous low-dose ketamine and epidural morphine in gastrectomy: a randomized double-blind study. Anesthesiology. 2000 Jun;92(6):1624-30. doi: 10.1097/00000542-200006000-00020. PMID 10839912
- [Background] Kararmaz A, Kaya S, Karaman H, Turhanoglu S, Ozyilmaz MA. Intraoperative intravenous ketamine in combination with epidural analgesia: postoperative analgesia after renal surgery. Anesth Analg. 2003 Oct;97(4):1092-1096. doi: 10.1213/01.ANE.0000080205.24285.36. PMID 14500163
- [Background] Ilkjaer S, Nikolajsen L, Hansen TM, Wernberg M, Brennum J, Dahl JB. Effect of i.v. ketamine in combination with epidural bupivacaine or epidural morphine on postoperative pain and wound tenderness after renal surgery. Br J Anaesth. 1998 Nov;81(5):707-12. doi: 10.1093/bja/81.5.707. PMID 10193280
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Ngan Kee WD, Khaw KS, Ma ML, Mainland PA, Gin T. Postoperative analgesic requirement after cesarean section: a comparison of anesthetic induction with ketamine or thiopental. Anesth Analg. 1997 Dec;85(6):1294-8. doi: 10.1097/00000539-199712000-00021. PMID 9390597
- [Background] Kashefi P. The benefits of intraoperative small-dose ketamine on postoperative pain after cesarean section. Anesthesiology 2006;104, Supp 1.
- [Background] Sen S, Ozmert G, Aydin ON, Baran N, Caliskan E. The persisting analgesic effect of low-dose intravenous ketamine after spinal anaesthesia for caesarean section. Eur J Anaesthesiol. 2005 Jul;22(7):518-23. doi: 10.1017/s026502150500089x. PMID 16045141
- [Background] Downing JW, Mahomedy MC, Jeal DE, Allen PJ. Anaesthesia for Caesarean section with ketamine. Anaesthesia. 1976 Sep;31(7):883-92. doi: 10.1111/j.1365-2044.1976.tb11899.x. PMID 9839
- [Background] Dich-Nielsen J, Holasek J. Ketamine as induction agent for caesarean section. Acta Anaesthesiol Scand. 1982 Apr;26(2):139-42. doi: 10.1111/j.1399-6576.1982.tb01741.x. PMID 7102236
- [Background] Maduska AL, Hajghassemali M. Arterial blood gases in mothers and infants during ketamine anesthesia for vaginal delivery. Anesth Analg. 1978 Jan-Feb;57(1):121-3. doi: 10.1213/00000539-197801000-00026. No abstract available. PMID 24371
- [Background] Bar-Oz B, Bulkowstein M, Benyamini L, Greenberg R, Soriano I, Zimmerman D, Bortnik O, Berkovitch M. Use of antibiotic and analgesic drugs during lactation. Drug Saf. 2003;26(13):925-35. doi: 10.2165/00002018-200326130-00002. PMID 14583068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at Prentice Women's Hospital between August 2006 and November 2006.
Pre-assignment Details: 188 subjects were recruited for the study. 5 subjects in the ketamine group and 3 in the saline group were excluded after randomization but before study drug administration.
Period: Overall Study
Arm/Group | Ketamine | Placebo
Started | 94 | 94
Completed | 85 | 89
Not Completed | 9 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — decision for postpartum tubal ligation | 3 | 1
Not completed — spinal anesthetic protocal violation | 1 | 1
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — No toradol due to hemmorhage or allergy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Placebo | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 94 | 188
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (3) | 34 (3) | 34 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 94 | 188
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 90 | 86 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 71 | 76 | 147
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  United States | 94 | 94 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Requiring Supplemental Analgesia in the First 24 Hours Following Cesarean Delivery
Description: Request for oral hydrocodone/acetaminophen for pain not controlled by around the clock non-steroidal antiflammatory drugs in the first 24 hours following cesarean delivery.
Time Frame: 24 hours
Population: Analysis was performed per protocol
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
participants | 64 | 66
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Sample size was determined assuming an incidence of breakthrough pain of 75% and an absolute difference between groups of -20 to +15%. This rate of request for analgesia in the first 24 h was based on data from a parallel study utilizing the same multimodal postoperative pain regimen for cesarean delivery. Group sample sizes of 90 achieve 80% power to detect this difference using the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.05; Test type: Superiority or Other; p = 0.86, Fisher Exact

2. Secondary Outcome: Verbal Pain Scores (0 to 10) at First Analgesia Request
Description: Numeric rating of pain scores (NRS) scale (0 to 10) at time of supplemental analgesia request. Zero is no pain and 10 is worst pain imaginable.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
Scores on a scale | 3 [2 to 4] | 4 [2 to 5]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Cumulative Hydrocodone/Acetaminophen for Supplemental Analgesia to Treat Breakthrough Pain
Description: Cumulative hydrocodone/acetaminophen for supplemental analgesia to treat breakthrough pain for 72 hours following cesarean delivery
Time Frame: 72 hours
Population: Analysis was per protocol
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
tablets | 10 [6 to 14] | 9 [5 to 12]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Postoperative Nausea
Description: Number of subjects reporting nausea in first 24 hours following cesarean delivery
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
participants | 27 | 30
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.87, Fisher Exact

5. Secondary Outcome: Postoperative Vomiting
Description: Number of subjects that vomited in the first 24 hours following cesarean delivery
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
participants | 13 | 13
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.90, Fisher Exact

6. Secondary Outcome: Postperative Pruritus
Description: Number of subjects with pruritus in the first 24 hours following cesarean delivery
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
participants | 12 | 19
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.24, Fisher Exact

7. Secondary Outcome: Disturbing Dreams
Description: Number of subject reporting disturbing dreams at 72 hours post cesarean delivery
Time Frame: 72 hours
Measure: Number; unit: participants
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
participants | 0 | 0
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 1.0, Fisher Exact

8. Post Hoc Outcome: Pain Score (0-10) at 2 Weeks Following Cesarean Delivery
Description: Numeric rating for pain score (0 to 10) reported at 2 weeks following cesarean delivery. Zero is no pain and 10 is worst pain imaginable.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 85 | 89
Scores on a scale | 2 [1 to 3] | 2.6 [1 to 4]
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority or Other; p = 0.02, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to -0.09]

ADVERSE EVENTS:
Arm/Group | Ketamine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/89
Other Adverse Events (participants affected / at risk) | 30/85 | 7/89
OTHER ADVERSE EVENTS (reported when occurring in more than 0.01% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=85) | Placebo (N=89)
Spontaneous complaint of psycho-mimetic reaction (Psychiatric disorders) | 30 (30) | 7 (7) — Spontaneous complaint of psycho-mimetic reaction (feeling clumsy or weird feeling) reported by subject 5 minutes after administration of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes